CLINICAL TRIAL: NCT02946983
Title: Influence of Intragastric Fructose Infusion on Behavioural and Neural Responses to Negative Emotion Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: S57996
Record Dates: First submitted 2016-05-12; First posted 2016-10-27 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Fructose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fructose - Neutral emotion condition (Active Comparator): Intragastric infusion of fructose with neutral emotion induction
  Interventions: Other: Fructose
- Fructose - Sad emotion condition (Active Comparator): Intragastric infusion of fructose with sad emotion induction
  Interventions: Other: Fructose
- Placebo - Neutral emotion condition (Placebo Comparator): Intragastric infusion of distilled water with neutral emotion induction
  Interventions: Other: Control
- Placebo - Sad emotion condition (Placebo Comparator): Intragastric infusion of distilled water with sad emotion induction
  Interventions: Other: Control

INTERVENTIONS:
Other: Fructose — Intragastric administration of fructose (25g dissolved in 250ml distilled water)
  Arms: Fructose - Neutral emotion condition; Fructose - Sad emotion condition
Other: Control — Intragastric administration of distilled water
  Arms: Placebo - Neutral emotion condition; Placebo - Sad emotion condition

SUMMARY:
The investigators will test whether a subliminal, intragastric dose of fructose is able to influence the emotional state at the behavioural and neural level, as has been previously shown for fatty acids. They will also examine the potential involvement of gut peptide release. Based on previous research using fatty acids, an attenuating effect of fructose compared to placebo on the induced negative emotional state is hypothesized at the self-report as well as the brain level.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (N=15)
* Male and female
* Age 18 - 60
* Body Mass Index (BMI) of 20 - 25 kg/m2
* Stable body weight for at least 3 months prior to the start of the study

Exclusion Criteria:

* Abdominal or thoracic surgery. Exception: appendectomy
* Gastrointestinal, endocrine or neurological diseases. Exception: IBS if the participant will be recruited in the patient group
* Cardiovascular, respiratory, renal or urinary diseases
* Hypertension
* Food or drug allergies
* Anemia
* Eating disorders
* Psychotic disorders
* Depressive disorders
* Emotional and/or restraint eating
* No medication on a regular basis, exception: oral contraception
* No history of cannabis use or any other drug of abuse for at least 12 months prior to the study
* Alcohol abuse (more than 21 units of alcohol for men, more than 14 units for woman per week)
* Conditions that can interfere with functional magnetic resonance imaging (fMRI), e.g. cochlear implants, metal fragments or metal implants in the body, pacemaker, neural stimulator, …
* Pregnant or breastfeeding women
* Claustrophobia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Functional brain images | From the start of the study until the endpoint of the study, with a total duration of 50 minutes
  Changes in brain responses after administration of our test solution compared to baseline will be assessed via functional magnetic resonance imaging

SECONDARY OUTCOMES:
Hunger scores | every 10 minutes since the scan starts until 40 minutes after the start of the scan
  The hunger scores will be taken every 10 minutes since the scan starts via a 10 cm visual analogue scale.
Mood assessment via the Self Assessment Manikin questionnaire | every 10 minutes since the scan starts until 40 minutes after the start of the scan
  Mood will be assessed every 10 minutes since the scan starts via the Self Assessment Manikin questionnaire
Gut hormone levels | every 10 minutes since the scan starts until 40 minutes after the start of the scan
  Peripheral blood samples will be taken every 10 min since the scan starts until the endpoint of the study to measure gut hormones (motilin, ghrelin, CCK, PYY, GLP-1) by radioimmuno-assay.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Prof, Principal Investigator — University of Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iven J, Biesiekierski JR, Zhao D, Tack J, Van Oudenhove L. Intragastric fructose administration interacts with emotional state in homeostatic and hedonic brain regions. Nutr Neurosci. 2022 Mar;25(3):581-592. doi: 10.1080/1028415X.2020.1781326. Epub 2020 Jun 19. PMID 32558624